CLINICAL TRIAL: NCT01370434
Title: Two Cycles of Pad Combination (Ps-341/Bortezomib, Adriamycin, and Dexamethasone) Followed by Autologous Hematopoietic Cell Transplantation in Newly Diagnosed Multiple Myeloma Patients
Brief Title: Two Cycles of PAD Combination by AHCT in MM
Acronym: PADinMM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: AMC, Asan Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-34
Record Dates: First submitted 2011-05-16; First posted 2011-06-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Multiple Myeloma
Keywords: MM
MeSH Terms: conditions — Multiple Myeloma | interventions — Vincristine; Doxorubicin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VAD combination (No Intervention): * vincristine 0.4mg iv on D1-4
  * doxorubicin 9mg/m2 iv on D1-4
  * dexamethasone 40mg/d po on D1-4,9-12,17-20
  * Many physicians use vincristine, doxorubicin, and dexamethasone (VAD) for three to four months as induction therapy (Alexandrian et al, 1990). VAD produces partial response (PR) in about 50% patients, with complete response (CR) observed in 5%-10% patients (Kyle et al, 2004).
  Interventions: Drug: PAD combination

INTERVENTIONS:
Drug: PAD combination — * Bortezomib 1.3 mg/m2/d iv on D 1, 4, 8, 11
  * Doxorubicin 9 mg/m2/d iv on D 1-4
  * Dexamethasone 40mg/d po or iv on D1-4, 8-11
  Other Names: -vincristine; -doxorubicin; -dexamethasone

SUMMARY:
Based the proven efficacy and the ability to induce rapid response of various combinations of bortezomib including PAD combination in refractory and newly diagnosed patients with Multiple Myeloma, the investigators intend to investigate the efficacy of 2 cycles of PAD combination (Ps-341/Bortezomib, Adriamycin, and Dexamethasone) and to examine the feasibility of harvesting G-CSF mobilized PBSC and performing early AHCT after 2 cycles of PAD.

DETAILED DESCRIPTION:
1.PAD combination chemotherapy

* Bortezomib 1.3 mg/m2 will be given by intravenous bolus injection on days 1, 4, 8, 11 of each cycle. Oral or intravenous dexamethasone 40 mg will be administered on days 1-4 and 8-11 with doxorubicin 9 mg/m2 by intravenous bolus on days 1-4 of each cycle. The cycle will be repeated every 3 weeks. A total of 2 cycles is planed before AHCT.
* For mobilization, G-CSF 10ug/kg/d alone will be given by subcutaneous injection from day 12 of the second PAD cycle until completion of harvesting.

Melphalan 100 mg/m2/day will be administered on day -3 and day -2 for high-dose chemotherapy.

-Maintenance :Thalidomide 100 - 200 mg/d for 2 years

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed symptomatic MM (see Appendix I)
* Patients should be eligible for AHCT.
* Patients should have measurable serum or urine paraprotein.
* The performance status of the patients should be 70 or over by Karnofsky performance scale
* Adequate hepatic and renal function: serum bilirubin < 1.5 x the upper limit of normal (ULN), serum alanine aminotransferase (ALT)/aspartate aminotransaminase (AST) values < 2.5 x ULN, serum creatinine < 1.5 x ULN
* Adequate cardiac function: ejection fraction > 40% by echocardiogram or radionuclide heart scan

Exclusion Criteria:

* prior chemotherapy for myeloma except 4 days of dexamethasone up to 40 mg per day or localized radiotherapy or plasmapheresis for the treatment of clinically significant hyperviscosity syndrome
* have a peripheral neuropathy of grade 2 or more within 14 days of enrollment.
* significant infection

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
response rates and toxicities. | 2.5 years
  To investigate the effectiveness of bortezomib, doxorubicin and dexamethasone (PAD) combination therapy in the treatment of previously untreated patients with multiple myeloma who are eligible for autologous hematopoietic cell transplantation (AHCT). The effectiveness will be evaluated in terms of response, response rates, and toxicities.

SECONDARY OUTCOMES:
hematologic recovery | 2.5 years
  To evaluate the feasibility of harvesting peripheral blood stem cells (PBSC) and performing AHCT after 2 cycles of PAD in newly diagnosed MM. Cell counts of harvested PBSC and hematologic recovery after AHCT will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hee Lee, professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Asanbyeongwon-gil, Songpa-gu, South Korea

REFERENCES:
- See also: Two Cycles of PAD Combination by AHCT in MM (PADinMM) — http://www.google.co.kr